CLINICAL TRIAL: NCT02245074
Title: Non Invasive Evaluation of Bronchial Inflammation in Infants : a Study of the Sputum Cellularity After Hypertonic Saline Induction
Acronym: CYTOASTHME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2009/056/HP; 2009- A00774-53 (Other: AFSSAPS)
Record Dates: First submitted 2010-10-15; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Infantile Asthma
Keywords: Infantile asthma; Induced sputum; Phenotypes; Eosinophils; Neutrophils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acute exacerbation (Other): Cell profiles Analysis after sputum induction in infants with Acute exacerbation
  Interventions: Other: Sputum induction
- Uncontrolled asthma (Other): Cell profiles Analysis after sputum induction in infants with Uncontrolled asthma
  Interventions: Other: Sputum induction
- controlled asthma (Other): Cell profiles Analysis after sputum induction in infants controlled asthma
  Interventions: Other: Sputum induction

INTERVENTIONS:
Other: Sputum induction — The sputum induction will be performed by repeated nebulizations of 3% saline hypertonic solution. Cellularity and cell profiles were analysed as previously recommended.

SUMMARY:
* Background: Infantile asthma is composed of various phenotypes, however the definition is still based on the clinics. Namely, the infants could be classified as transitory, peristent or late and persistent asthma. Some risk factors for the persistent asthma phenotype are recognized as atopy. However all peristent asthma are not related to atopy. Regarding the pathophysiology, little is known on airways inflammation in these infants, and the current data are mostly based on the BAL analyses, or on biopsies. Consequently, BLA and biopsies should be justified by the need of an indicated fiberbronchoscopy, and therefore limited to severe infantile asthma. Airway secretion could be also collected after hypertonic saline induction and chest physiotherapy. This method has been validated in the children, but has not in the younger.
* Aim : Analyses of cell profiles regarding the severity of infantile asthma.
* Methods : This descriptive study compared 3 groups of infants, the first with acute exacerbation, the second with uncontrolled asthma and the third with controlled asthma. Accounting 25% of failure, the number of 40 infants per groups has been calculated. The sputum induction will be performed by repeated nebulizations of 3% saline hypertonic solution. Cellularity and cell profiles were analysed as previously recommended. Safety will be evaluated.
* Inclusion criteria : Any infants suffering of infantile asthma (at least 3 episodes of wheezing during the 2 first years of life), aged between 6-12months.Asthma control was evaluated on the last 4 weeks, allowing to classify the infants . Control asthma was aimed when neither exacerbation nor persistent symptoms were observed. Uncontrolled asthma was defined whether the infant presented any symptoms during the last 4 weeks. Exacerbation was defined as any acute symptoms, as cough, dyspnoea or wheezing.
* Feasibility : A preliminary study has been presented in the Vienna ERS congress.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 36 mo.
* Ambulatory or hospitalized.
* With %SaO2 ³ 95%
* Parents information and non-opposition from the parents

Exclusion Criteria:

* Any underlying chronic disease
* Been given oral corticosteroid during the last four weeks
* Known adverse events with nebulized saline solution
* With cold during the 4 last weeks for the controled group.
* With %SaO2 < 95%

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Cell profiles Analysis regarding the severity of asthma as defined above. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Christophe MARGUET, Professor, Principal Investigator — University Hospital, Rouen
Locations (1):
- Pediatric Department, Rouen, France